CLINICAL TRIAL: NCT01365637
Title: A Double Blind (3rd Party Open) Randomized, Placebo Controlled, Parallel Group Multiple Dose Escalation Study To Investigate The Safety, Toleration And Pharmacokinetics Of PF-05089771 In Healthy Subjects.
Brief Title: The Safety and Tolerability of PF-05089771 Will be Investigated in Healthy Subjects Over a 14 Day Dosing Period.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3291002
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Pain
Keywords: safety; tolerability; pharmacokinetics; PF-05089771
MeSH Terms: conditions — Pain | interventions — PF-05089771

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 PF-05089771 or placebo (Experimental): Subjects will receive multiple doses of PF-05089771 or placebo twice daily to investigate the safety/tolerability and PK of PF-05089771. The PK of alternative formulations of PF-05089771 and the effect of food on PK may also be investigated.
  Interventions: Drug: PF-05089771
- Cohort 2 PF-05089771 or placebo (Experimental): Subjects will receive multiple doses of PF-05089771 or placebo twice daily to investigate the safety/tolerability and PK of PF-05089771. The PK of alternative formulations of PF-05089771 and the effect of food on PK may also be investigated.
  Interventions: Drug: PF-05089771
- Cohort 3 PF-05089771 or placebo (Experimental): Subjects will receive multiple doses of PF-05089771 or placebo either twice or thrice daily to investigate the safety/tolerability and PK of PF-05089771. The PK of alternative formulations of PF-05089771 and the effect of food on PK may also be investigated.
  Interventions: Drug: PF-05089771
- Cohort 4 PF-05089771 or placebo (Experimental): Subjects will receive multiple doses of PF-05089771 or placebo either twice or thrice daily to investigate the safety/tolerability and PK of PF-05089771. The PK of alternative formulations of PF-05089771 and the effect of food on PK may also be investigated.
  Interventions: Drug: PF-05089771

INTERVENTIONS:
Drug: PF-05089771 — PF-05089771 will be dosed as a suspension twice daily
  Arms: Cohort 1 PF-05089771 or placebo
Drug: PF-05089771 — PF-05089771 will be dosed as a suspension twice daily
  Arms: Cohort 2 PF-05089771 or placebo
Drug: PF-05089771 — PF-05089771 will be dosed as a suspension either twice or thrice daily
  Arms: Cohort 3 PF-05089771 or placebo
Drug: PF-05089771 — PF-05089771 will be dosed as a suspension either twice or thrice daily
  Arms: Cohort 4 PF-05089771 or placebo

SUMMARY:
The purpose of the study is primarily to determine the safety and toleration and pharmacokinetics of PF-05089771 following escalating multiple doses lasting for 14 days. Dosing will either be administered twice or three times daily. Secondary objectives will be to investigate the PK of an alternative formulation of PF-05089771 and the effect of food on the PK of PF-05089771.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects or female subjects of non-child bearing potential between the ages of 18 and 55 years, inclusive.

Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

An informed consent document signed and dated by the subject

Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (e.g., gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 21 drinks/week (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug within 60 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* 12-lead ECG demonstrating QTc >450 msec at screening.
* If QTc exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* Females of child bearing potential.
* Use of prescription or non-prescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements must be discontinued 28 days prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of 1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of PF-05089771 | Days 1-16
Maximum concentration (Cmax) for PF-05089771 in plasma (measured in ng/mL) | Days 1-16
Tmax = Time of maximum concentration of PF-05089771 in plasma (hr) | Days 1-16
AUCtau= Area under the curve from the time of dosing to the next dose (ng.hr/mL) | Days 1-16
Elimination half life (hr) = rate of elimination of PF-05089771 after the final dose | Days 14-16

SECONDARY OUTCOMES:
AUCinf = Area under the curve from the time of dosing extrapolated to infinity (ng.hr/mL) | Days 14-16

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3291002&StudyName=The%20safety%20and%20tolerability%20of%20PF-05089771%20will%20be%20investigated%20in%20healthy%20subjects%20over%20a%2014%20day%20dosing%20period.%20